CLINICAL TRIAL: NCT03511638
Title: A Study to Document the Safety and Effectiveness of a New OVD When Compared to a Control OVD
Brief Title: Bausch & Lomb Ophthalmic Viscosurgical Device (OVD) Dispersive (DVisc40)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S877
Record Dates: First submitted 2017-11-17; First posted 2018-04-30 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: a multicenter, controlled, randomized, monocular trial of Bausch & Lomb DVisc40 (test) OVD compared to the currently marketed Alcon VISCOAT® (control) OVD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Bausch & Lomb DVisc40 (Experimental): Ophthalmic viscosurgical device
  Interventions: Device: Bausch & Lomb DVisc40
- Alcon VISCOAT® (Active Comparator): Ophthalmic viscosurgical device
  Interventions: Device: Alcon VISCOAT®

INTERVENTIONS:
Device: Bausch & Lomb DVisc40 — Ophthalmic viscosurgical device
  Arms: Bausch & Lomb DVisc40
Device: Alcon VISCOAT® — Ophthalmic viscosurgical device
  Arms: Alcon VISCOAT®

SUMMARY:
A Study to Document the Safety and Effectiveness of a New OVD When Compared to a Control OVD

DETAILED DESCRIPTION:
This is a multicenter, controlled, randomized, monocular trial evaluating the safety and effectiveness of the Bausch & Lomb DVisc40 dispersive OVD compared to the Alcon VISCOAT® dispersive OVD when used in cataract surgery. Subjects will be randomized to one of the two treatment groups in a 1:1 ratio (DVisc40:VISCOAT®).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 45 years old and have a clinically documented diagnosis of age-related non-complicated cataract that is considered amenable to treatment with standard phacoemulsification cataract extraction and IOL implantation.

  2. The subject must have the capability to provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.

  3. The subject must be willing and able to return for all scheduled follow-up examinations through 90 days following surgery.

Study #877 Protocol DVisc40 28JUL2017 V1.0 CONFIDENTIAL Page 16 of 53 4. The subject must have clear intraocular media other than the cataract in the operative eye.

Exclusion Criteria:

* 1. The subject has participated in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.

  2. The subject has any corneal pathology (e.g., significant scarring, guttata, inflammation, edema, dystrophy, etc.) in the operative eye.

  3. The subject has anterior segment pathology likely to increase the risk of an adverse outcome for phacoemulsification cataract surgery (e.g., pseudoexfoliation syndrome, synechiae, iris atrophy, inadequate dilation, shallow anterior chamber, traumatic cataract, lens subluxation) in the operative eye.

  4. The subject has any condition which prevents reliable specular microscopy in the operative eye.

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Valeant Site 01, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bausch & Lomb DVisc40 | Alcon VISCOAT®
Started | 184 | 188
Completed | 182 | 187
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bausch & Lomb DVisc40 | Alcon VISCOAT® | Total
Number analyzed (Participants) | 184 | 188 | 372
Age, Continuous [Median (Full Range); unit: years] | 70.0 [47 to 86] | 69.0 [45 to 86] | 70.0 [45 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 120 | 231
  Male | 73 | 68 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 39 | 43 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 7 | 26
  White | 122 | 136 | 258
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 1
Study eye - right or left [Count of Participants; unit: Participants]
  Right Eye | 91 | 110 | 201
  Left Eye | 93 | 78 | 171

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Epithelial Cell Density (ECD)
Time Frame: Day 90
Population: Participants with epithelial cell density at baseline and Day 90 were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change in ECD
Arm/Group | Bausch & Lomb DVisc40 | Alcon VISCOAT®
Number analyzed (Participants) | 168 | 178
percentage change in ECD | -8.4 (12.19) | -6.8 (12.54)

2. Primary Outcome: Percentage of Participants With Postoperative Intraocular Pressure of at Least 30 mm Hg
Time Frame: 90 days
Measure: Number; unit: percentage of participants
Arm/Group | Bausch & Lomb DVisc40 | Alcon VISCOAT®
Number analyzed (Participants) | 184 | 188
percentage of participants | 17.4 | 20.3

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Bausch & Lomb DVisc40 | Alcon VISCOAT®
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/188
Serious Adverse Events (participants affected / at risk) | 1/184 | 4/188
Other Adverse Events (participants affected / at risk) | 48/184 | 51/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bausch & Lomb DVisc40 (N=184) | Alcon VISCOAT® (N=188)
Posterior capsule rupture (Eye disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bausch & Lomb DVisc40 (N=184) | Alcon VISCOAT® (N=188)
Punctate keratitis (Eye disorders) | 17 | 13
Intraocular pressure increased (Investigations) | 31 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03511638/Prot_SAP_000.pdf